CLINICAL TRIAL: NCT06947369
Title: The Effects of Education Given to Primiparous Pregnant Women Who Have Fear of Childbirth According to Joyce Travelbee's Human-to-Human Relationship Model on Fear of Childbirth, Readiness for Childbirth and Acceptance of the Maternal Role
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Funda Gul Bilgen, PhD Student, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/018
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Fear of Childbirth, Pregnant Woman; Healthy Pregnant Woman; Healt
Keywords: Primiparous pregnant, fear of childbirth,role of motherhood, Joyce Travelbee, childbirth readiness

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Within the scope of the research, the pregnant women in the experimental group will be given a training program based on Joyce Travelbee's human-to-human relations theory, one session per week for 30-45 minutes, for a total of five sessions.
  Interventions: Other: Experimental Group
- Control group (No Intervention): Within the scope of the research, no training will be given to the control group after the pretest is applied.

INTERVENTIONS:
Other: Experimental Group — Within the scope of the research, the pregnant women in the experimental group will be given a training program based on Joyce Travelbee's human-to-human relations theory, one session per week for 30-45 minutes, for a total of five sessions, while the control group will continue their routine follow-up.
  Arms: Experimental group

SUMMARY:
The research is planned as a randomised controlled experimental study. Research data will be collected between March-July 2025. The population of the study will consist of all pregnant women who come to Kilis Prof.Dr.Alaeddin Yavaşca State Hospital Gynaecology and Obstetrics Polyclinics. The sample of the study will consist of primiparous pregnant women who meet the research criteria and accept to participate in the study among the pregnant women who come to Kilis Prof.Dr.Alaeddin Yavaşca State Hospital Gynaecology and Obstetrics Polyclinics.

Data will be collected from primiparous pregnant women who meet the inclusion criteria and accept the study after being informed about the study by meeting the pregnant women who come to Kilis Prof.Dr.Alaeddin Yavaşca State Hospital Gynaecology and Obstetrics Outpatient Clinic before or after their outpatient examinations.

Data Collection Tools Personal Information Form, Wijma Birth Anticipation / Experience Scale A Version scale and Prenatal Self-Assessment Scale Dependent variables of the study: Wijma Birth Expectancy / Experience Questionnaire (W-DEQ) A Version and Prenatal Self-Assessment Scale subscales of acceptance of maternal role and readiness for childbirth scales. Independent variables of the study: Socio-demographic and obstetric characteristics of primiparous pregnant women

DETAILED DESCRIPTION:
3. METHODS AND TECHNIQUES Type and Time of the Study The study is planned as a randomised controlled experimental study.

Research data will be collected between March-July 2025. Hypotheses (H):

H0a: The training given to primiparous pregnant women with fear of childbirth according to Joyce Travelbee's Human Human Human Relationship Model does not affect fear of childbirth.

H1a: The training given to primiparous pregnant women with fear of childbirth according to Joyce Travelbee's Human Human Human Relationship Model affects fear of childbirth.

H0b: The education given to primiparous pregnant women experiencing fear of childbirth according to Joyce Travelbee's Human Human Human Relationship Model does not affect the level of birth readiness.

H1b: The education given to primiparous pregnant women with fear of childbirth according to Joyce Travelbee's Human Human Human Relationship Model affects the level of birth readiness.

H0c: The training given to primiparous pregnant women with fear of childbirth according to Joyce Travelbee's Human Human Human Relationship Model does not affect the acceptance of the maternal role.

H1c:The training given to primiparous pregnant women experiencing fear of childbirth according to Joyce Travelbee's Human-Human Relationship Model affects the acceptance of the maternal role. Ethical Aspects of the Study - Ethical approval was obtained from Hasan Kalyoncu University, Faculty of Health Sciences, Non-Interventional Research Ethics Committee for the conduct of the study - Written permissions were obtained from Kilis Prof.Dr.Alaeddin Yavaşca State Hospital and Kilis Provincial Health Directorate where the study will be conducted.

- Informed consent/voluntary consent form will be obtained from primiparous women participating in the study. With the informed consent form, the pregnant women will be informed in detail about the purpose of the education to be given to the pregnant women, the identity of the researcher, the information to be obtained from the pregnant women will be kept confidential and will not be shared, and where and how the information obtained will be used. Pregnant women will also be informed that they can withdraw from the study at any time. - Permission for use was obtained from the authors of the validity and reliability scales used in the study.

The Universe and Sample of the Study The universe of the study will consist of all pregnant women who come to the Gynecology and Obstetrics Clinics of Kilis Prof. Dr. Alaeddin Yavaşca State Hospital. The sample of the study will consist of primiparous pregnant women who meet the research criteria and accept to participate in the study among the pregnant women who come to the Gynecology and Obstetrics Clinics of Kilis Prof. Dr. Alaeddin Yavaşca State Hospital.

When calculating the sample size in randomized controlled experimental studies, the difference between the groups refers to the absolute difference between the groups compared in clinical studies. The d / EB (Effect Size) value used to determine the sample size in the study was taken from the standardized effect size found in similar studies by scanning the literature (Demirci & Şimşek, 2018). The G*Power version 3.1.9.7 program was used to calculate the size and power value of the research sample. The study conducted by Demirci and Şimşek was taken as a reference in the sample size calculation (Demirci & Şimşek, 2018). According to the G Power analysis, with a 5% margin of error, 90% power (representing the universe) and an effect size of 0.884, a total of 28 and 56 were calculated in both groups. Considering the patients who would not continue the study and who could withdraw from the study during the study, it was decided to add 7 people to each group in terms of possible sample loss, making 35 for each group and 70 people in total.

Criteria for participation in the study

1. The pregnant woman's first pregnancy.
2. A mid-level or above score on the Wijma Childbirth Expectation/Experience Scale Version A scale.
3. The pregnant woman's being between 28-40 weeks of gestation (third trimester).
4. The pregnant woman's not having a chronic health problem.
5. The pregnant woman having a single fetus.
6. The pregnant woman not having received infertility treatment.
7. The pregnant woman not having received a psychiatric diagnosis.
8. The pregnant woman does not have a high-risk pregnancy (placenta previa, antepartum hemorrhage history, membrane rupture, preeclampsia, hypertension, diabetes or other medical conditions, intrauterine growth retardation, fetal anomalies or any contraindication to normal vaginal delivery, drug or alcohol addiction).
9. The pregnant woman agrees to participate in the study. Exclusion Criteria from the Study

1. Those who do not volunteer to participate in the study 2. Those who do not speak Turkish 3. Those who are illiterate or have difficulty communicating 4. Those who do not meet the study criteria Exclusion criteria from the study Women who accept the application but later decide not to continue the application or do not continue Randomization and Blinding In order to ensure equal distribution between the groups, the participants to be included in the intervention and control groups will be determined by randomization using the simple randomization method (https://www.randomizer.org/) (Kanık, Taşdelen, & Erdoğan, 2011). Randomization will be performed by a person independent of the study.

The study was planned as a one-way blinded study because the women in the study did not know which experimental or control group they were in, but the researcher did. After randomization, statistical analysis of independent variables such as age, marriage duration, education status and employment status of the intervention and control groups will be performed to verify the homogeneity of the groups.

Data Collection and Data Analysis Data will be collected from primiparous pregnant women who meet the criteria for inclusion in the study and accept the study after being informed about the study by meeting with the pregnant women who come to Kilis Prof. Dr. Alaeddin Yavaşca State Hospital Gynecology and Obstetrics Clinic before or after their outpatient clinic examinations.

All pregnant women who accept to participate in the study will be informed about how the study will proceed, that participation in the study is based on volunteering, the risks of the study, the possibility of refusing to participate in the study and withdrawing from the study at any time, and detailed informed consent forms will be signed by each pregnant woman.

Data Analysis The analysis of the data obtained from the study will be carried out in the SPSS 25 program. Categorical measurements will be stated as percentages. Mean and standard deviation values will be used in the descriptive statistics of the data. Whether the variables provide normal distribution will be measured with the Kolmogorov Simirnov/Shapiro-Wilk test. Parametric or nonparametric tests will be used depending on whether the data show normal distribution or not. Student t test will be used for comparing variables that follow a normal distribution between groups, and Mann Whitney U test will be used for variables that do not follow a normal distribution. Kurskall-Wallis H test will be applied to find the difference between three or more categorical variables. Correlation analysis will be performed to reveal the relationship between dependent variables. In addition, Wilcoxon test will be performed for the test of the difference between two different measurement times obtained from the same individuals. Regression tests will be used to determine the effectiveness of the training.

Data Collection Tools Personal Information Form, Wijma Birth Expectation/Experience Scale Version A scale and Prenatal Self-Assessment Scale Personal Information Form: The data collection tool prepared in line with the literature consists of a total of 32 questions (Aslan & Bıyık, 2020; Demir, 2023; Esenkaya & Gölbaşı, 2024). The content of the form includes the socio-demographic characteristics and obstetric information of pregnant women (Appendix-2).

Wijma Birth Expectation/Experience Scale (W-DEQ) Version A: It was developed by Wijma and colleagues in 1998 to determine the fear and stress of childbirth in pregnant women, and its validity and reliability in Turkish were performed by Körükçü and colleagues in 2012. W-DEQ version A is a 6-point Likert-type scale consisting of 33 items. The minimum score on the scale is 0, and the maximum score is 165. The negatively loaded questions in the scale (2, 3, 6, 7, 8, 11, 12, 15, 19, 20, 24, 25, 27, 31) are calculated by reversing. A high score indicates a high level of fear of childbirth. - W-DEQ score ≤ 37 indicates mild level,

* W-DEQ score = 38-65 indicates moderate level,
* W-DEQ score = 66-84 indicates severe level,
* W-DEQ score ≥ 85 indicates clinical level fear. The cut-off point is 85. A score of 85 and above indicates clinical level fear of childbirth. The Cronbach Alpha value of the scale was found to be 0.88 for primiparous pregnant women, 0.90 for multiparous pregnant women and 0.89 for the total group (Körükçü et al., 2012). (Appendix-3) Prenatal Self-Assessment Scale (PSS): The scale, which was developed by Lederman in 1979 to evaluate the adaptation of women to motherhood in the prenatal period, was evaluated for validity and reliability in Turkey by Beydağ and Mete in 2006 (Beydağ & Mete, 2008). In this study, the internal consistency coefficient of the scale was found to be high (α=0.81), and the internal consistency reliability coefficients of the subgroups were found to be between 0.72 and 0.85. PKDÖ is a 79-item, 4-point Likert-type scale with 7 sub-dimensions (thoughts about her own and her baby's health, acceptance of pregnancy, acceptance of the role of motherhood, readiness for birth, fear of birth, status of her relationship with her own mother, and status of her relationship with her husband). Each sub-scale has 10-15 items.

Each item in the scale is scored on a 4-point scale (4: Describes very much, 3: Partially describes, 2: Somewhat describes, 1: Does not describe at all). For reverse items (1, 2, 3, 4, 6, 7, 8, 10, 11, 12, 14, 15, 18, 19,20, 21, 22, 23, 24, 25, 26, 28, 31, 32, 33, 35, 37, 38, 40, 47, 48, 49, 50, 53, 55, 56, 59,60, 61, 70, 71, 72, 73, 74, 75, 78, 79), scoring is done in the opposite way. The minimum score for the entire scale is 79 and the maximum score is 316. Low scores indicate high adaptation to pregnancy, while high scores indicate low adaptation to pregnancy.

Approval was obtained from the scale authors regarding the suitability of using the subscales of the Prenatal Self-Assessment Questionnaire (PSQQ) separately.

Dependent variables of the study: Wijma Birth Expectation/Experience Questionnaire (W-DEQ) Version A and Prenatal Self-Assessment Questionnaire subscales Acceptance of the maternal role and Birth readiness scales.

Independent variables of the study: Socio-demographic and obstetric characteristics of primiparous pregnant women Data Collection Process Step 1: Among the pregnant women who come to the outpatient clinic examination, those who are suitable according to the study criteria and those who accept the study will first fill out the Personal Information Form and Wijma Birth Expectation/Experience Questionnaire Version A scale to determine their compliance with the research criteria. Pregnant women who score at the middle level and above on this scale will be selected. Contact information will be obtained from pregnant women who accept the study. In order to ensure homogeneity within the group, Experimental and Control groups will be created through randomization. The subscales of the Prenatal Self-Assessment Scale, which are the Pre-test data collection tools, Readiness for Birth and Acceptance of the Maternal Role scales, will be applied to the experimental and control groups.

Phase 2: Within the scope of the research, the training program based on Joyce Travelbee's human-to-human relations theory will be applied to the pregnant women in the experimental group for a total of five sessions, one session per week for 30-45 minutes, while the control group will continue its routine follow-up.

Phase 3: After the completion of the training program, the Wijma Birth Expectation/Experience Scale Version A scale, the Prenatal Self-Assessment Scale subscales, Readiness for Birth and Acceptance of the Maternal Role scales will be applied to the experimental and control groups to obtain post-test data to determine the change in primiparous pregnant women.

The content of the training program; The topics of "Formation-physiology of pregnancy, Signs-stages of the beginning of labor, Defining fear of childbirth, Explanation of types of childbirth, What to do in preparation for childbirth, Baby care" will be prepared within the framework of literature. Expert opinion will be sought to evaluate the suitability of the training content. Training content will be adjusted in line with the feedback from experts.

ELIGIBILITY:
Inclusion Criteria:1. The pregnant woman's first pregnancy. 2. A mid-level or above score on the Wijma Childbirth Expectation/Experience Scale Version A.

3. The pregnant woman is between 28-40 weeks of gestation (third trimester). 4. The pregnant woman does not have a chronic health problem. 5. The pregnant woman has a single fetus. 6. The pregnant woman has not received infertility treatment. 7. The pregnant woman has not received a psychiatric diagnosis. 8. The pregnant woman does not have a high-risk pregnancy. 9. The pregnant woman's acceptance to participate in the study.

Exclusion Criteria:1. Not willing to participate in the study 2. Not speaking Turkish 3. Illiterate, having communication difficulties 4. Not meeting the study criteria

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Primiparous pregnant women
Enrollment: 70 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Information about the physiology of pregnancy and the pregnancy process | 1 week after the pretest was administered
  * Briefly introducing herself
  * How she felt when she learned she was pregnant
  * How she perceived and adapted to pregnancy
  * Questioning the pregnancy process and providing information on the subject

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr.Ümran SEVİL, Study Director — Hasan Kalyoncu University
Locations (1):
- Kilis Prof.Dr.Alaeddin Yavaşca State Hospital, Kilis, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No